CLINICAL TRIAL: NCT05503030
Title: A Prospective, Observational Study on the Correlations Between Change in Lung Function and Change in Cough and Dyspnoea in Patients With Connective Tissue Disease-associated Progressive Fibrosing INTErstitial luNg diseaSE (CTD Associated PF-ILD) Treated With Nintedanib. The "INTENSE" Study
Brief Title: Correlation Between Changes in Lung Function and Changes in Cough and Dyspnoea in Nintedanib-treated Connective Tissue Disease Interstitial Lung Disease (CTD-ILD) Patients
Status: Terminated | Type: Observational
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1199-0501
Record Dates: First submitted 2022-08-15; First posted 2022-08-16 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Lung Diseases, Interstitial
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — nintedanib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Nintedanib for CTD-associated PF-ILD patients in Greece: Connective Tissue Disease (CTD)-associated Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
  Interventions: Drug: Nintedanib

INTERVENTIONS:
Drug: Nintedanib — Nintedanib

SUMMARY:
The aim of this study is to identify correlations between change from the baseline at Month 24 in Forced Vital Capacity (FVC) (% predicted and mL) and change from the baseline at Month 24 in cough or dyspnoea scores [points] as measured in the living with pulmonary fibrosis questionnaire (L-PF) over 24 months of nintedanib treatment in patients with connective tissues disease-associated progressive fibrosing interstitial lung disease (CTD associated PF-ILD) under routine clinical practice conditions in Greece.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years with a confirmed physician diagnosis of connective tissue disease (CTD) associated Progressive Fibrosing Interstitial Lung Disease (PF-ILD)
* Have been prescribed nintedanib according to the local Summary of Product Characteristics (SmPC) and clinical judgment. Therapy with nintedanib must have been started for clinical reasons independently from the intended patient enrolment into the study at a maximum of 15 days before enrolment into the trial.

Exclusion Criteria:

* Patients currently receiving treatment with any investigational drug/device/intervention or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with nintedanib
* Patients at baseline with a known condition or reason that will result in withdrawal from the study before the 24-month time point
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with physician-diagnosed interstitial lung disease (ILD) must fulfil at least one of the following criteria for progressive fibrosing (PF)-ILD within the previous period and up to two years before the screening, despite standard treatment to treat ILD:
  * Clinically significant decline in forced vital capacity (FVC) percentage (%) predicted based on a relative decline of ≥ 10%
  * The marginal decline in FVC % predicted based on a relative decline of ≥ 5-< 10% combined with worsening respiratory symptoms
  * The marginal decline in FVC % predicted based on a relative decline of ≥ 5-< 10% combined with increasing extent of fibrotic changes on chest imaging
  * Worsening of respiratory symptoms as well as increasing extent of fibrotic changes on chest imaging All patients will need to be treatment naïve concerning antifibrotic treatments (i.e., nintedanib or pirfenidone) before initiating nintedanib. Enrolment period will be 24 months, and each participant will be observed for 24 months.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Correlation between change from baseline at Month 24 in forced vital capacity (FVC) [percentage (%) predicted] and change from baseline at Month 24 in dyspnoea symptom score [points] | At baseline and at month 24
  The "living with pulmonary fibrosis" (L-PF) questionnaire for dyspnea/cough symptom score consists of 44 items divided into two modules: Symptoms (23 items) and Impacts (21 items). The Symptoms module assesses shortness of breath (dyspnea), cough and fatigue over the last 24 hours. The Impacts module assesses multiple aspects of health related quality of life (HRQoL) over the last 7 days. Symptoms and Impacts scores are used to calculate a total score.
  Items in both modules have response options on a five-option numeric rating score with an anchor of 0 "Not at all" to 4 "Extremely". Overall scores range from 0 to 100, with higher numbers indicating a greater impairment.
Correlation between change from baseline at Month 24 in forced vital capacity (FVC) [% predicted] and change from baseline at Month 24 in cough symptom score [points] | At baseline and at month 24

SECONDARY OUTCOMES:
Correlation between the change from baseline at Month 24 in forced vital capacity (FVC) [milliLitres (mL)] and change from baseline at Month 24 in dyspnoea symptom score [points] | At baseline and at month 24
Correlation between change from baseline at Month 24 in FVC [mL] and change from baseline at Month 24 in cough symptom score [points] | At baseline and at month 24
Correlation between baseline FVC [% pred] and change in dyspnoea symptom score [points] from baseline at month 24 | At baseline and at month 24
Correlation between baseline FVC [% pred] and change in cough symptom score [points] from baseline at month 24 | At baseline and at month 24
Absolute change from baseline in FVC [% pred] at month 24 | At baseline and at month 24
Absolute change from baseline in FVC [mL] at month 24 | At baseline and at month 24
Absolute change from baseline in Living with Pulmonary Fibrosis (L-PF) dyspnoea symptom score [points] at month 24 | At baseline and at month 24
Absolute change from baseline in L-PF cough symptom score [points] at month 24 | At baseline and at month 24
Change in total L-PF score [points] from baseline at month 24, or the end of the observation | At baseline and up to 24 months

CONTACTS AND LOCATIONS:
Locations (17):
- Greece (17):
  - Private physician, Athens
  - "G. Gennimatas" General Hospital of Athens, Athens
  - "Ippokration" General Hospital of Athens, Athens
  - "Laiko" General Hospital of Athens, Athens
  - "ATTIKON" University General Hospital, Athens
  - "KAT" General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion
  - Private physician, Ioannina
  - University General Hospital of Ioannina, Ioannina
  - Private physician, Larissa
  - University General Hospital of Larisa, Larissa
  - Private physician, Nea Smirni, Athens
  - Private physician, Pátrai
  - University General Hospital of Patra, Pátrai
  - Private physician, Thessaloniki
  - "Hippokration" General Hospital of Thessaloniki, Thessaloniki
  - "G. Papanikolaou" General University of Thessaloniki, Thessaloniki

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'.
  For study data - 1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com